CLINICAL TRIAL: NCT05038358
Title: Tumor Immune Microenvironment Involvement in Colorectal Cancer Chemoresistance Mechanisms: a Patient-derived Tumoroids Prospective Collection From Systemic Treatment Naive Tumors
Brief Title: Tumor Immune Microenvironment Involvement in Colorectal Cancer Chemoresistance Mechanisms
Acronym: CRC-ORGA2
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-A00793-38
Record Dates: First submitted 2021-08-31; First posted 2021-09-09 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Primary Tumor; Colon Tumor
Keywords: Organoid collection from fresh human primary colonic tumor tissue
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Colorectal cancer is the third most common cancer worldwide and its progression-free survival is still low, around 10 months. Thirthy to 50% of patients do not respond to chemotherapy upon initiation of treatment, suggesting that early development of chemoresistance mechanisms remains a major challenge. In order to better characterize these mechanisms, the aim is to develop a model of tumoroids derived from patients with a colorectal tumors prior to any systemic anti cancer treatment. This project will both allow us to study the role of the immunological microenvironment in chemoresistance and identify new predictive markers of tumor response. It will then serve to develop innovative personalized medicine strategies by targeting the newly identified mechanisms. This study should in fine help to improve the cancer patient's care.

ELIGIBILITY:
Inclusion Criteria:

* Male and female over 18 years old.
* Managed at the CHUGA for a colorectal adenocarcinoma
* With an indication for immediate surgical resection as part of the care.
* Patient naive from neo-adjuvant chemotherapy
* Patient did not object to the CRC-ORGA-2 study

Exclusion Criteria:

* Patients protected by law (pregnant or breastfeeding women, minors, patients under guardianship or trusteeship, persons deprived of their liberty or hospitalized under duress).
* Patients with positive HIV, HBV, HCV serology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: colorectal adenocarcinoma, naive from neo-adjuvant chemotherapy, indication of surgical resection
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-12-12 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of viable organoids for 60 days of culture maintenance. | 60 days of culture maintenance.

CONTACTS AND LOCATIONS:
Overall Officials: GAEL ROTH, MD, PHD, Principal Investigator — university hospital of Grenoble alpes
Locations (1):
- University Hospital of Grenoble Alpes, Grenoble, France